CLINICAL TRIAL: NCT02950233
Title: NMDA Antagonists and Steroids for the Prevention of Persisting Post-Surgical Pain After Thoracoscopic Surgeries: A Randomized Controlled, Factorial Design, International, Multicentre Pilot Study
Brief Title: Preventing pAIn With NMDA Antagonists - Steroids in Thoracoscopic lObectomy Procedures (PAIN-STOP) Pilot Trial
Acronym: PAIN-STOP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment was slower than expected and study drug reached expiry
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-001-PS
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Pain, Postoperative
Keywords: postoperative pain; VATS; activities of daily living; quality of life
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: We will randomize patients in a 1:1:1:1 fashion to receive; 1) NMDA active + dexamethasone placebo, 2) dexamethasone active + NMDA placebo, 3) NMDA active + dexamethasone active, and 4) NMDA placebo + dexamethasone placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, health care providers, data collectors, outcome adjudicators, and Investigators (e.g., Steering Committee Members) will all be blind to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NMDA active + Steroid placebo (Experimental): NMDA active: ketamine (0.5 mg/kg IV bolus pre-incision and 0.1 mg/kg/hr infusion postoperatively up to 24 hours) and oral memantine (5 mg BID [first week]; 10 mg BID [following three weeks]).
  Steroid placebo: two doses of normal saline; 25 mg given prior to starting surgery and 25 mg given on the morning of second postoperative day.
  Interventions: Drug: NMDA active; Drug: Steroid placebo
- Steroid active + NMDA placebo (Experimental): NMDA placebo: normal saline (IV bolus pre-incision and infusion postoperatively up to 24 hours) and oral matching placebo to memantine (one capsule BID [first week]; one capsule BID [following three weeks]).
  Steroid active: two doses of dexamethasone; 25 mg given prior to starting surgery and 25 mg given on the morning of second postoperative day.
  Interventions: Drug: Steroid active; Drug: NMDA placebo
- NMDA active + Steroid active (Experimental): NMDA active: ketamine (0.5 mg/kg IV bolus pre-incision and 0.1 mg/kg/hr infusion postoperatively up to 24 hours) and oral memantine (5 mg BID [first week]; 10 mg BID [following three weeks]).
  Steroid active: two doses of dexamethasone; 25 mg given prior to starting surgery and 25 mg given on the morning of second postoperative day.
  Interventions: Drug: NMDA active; Drug: Steroid active
- NMDA placebo + Steroid placebo (Placebo Comparator): NMDA placebo: normal saline (IV bolus pre-incision and infusion postoperatively up to 24 hours) and oral matching placebo to memantine (one capsule BID [first week]; one capsule BID [following three weeks]).
  Steroid placebo: two doses of normal saline; 25 mg given prior to starting surgery and 25 mg given on the morning of second postoperative day.
  Interventions: Drug: NMDA placebo; Drug: Steroid placebo

INTERVENTIONS:
Drug: NMDA active — NMDA active group will involve ketamine (0.5 mg/kg IV bolus pre-incision and 0.1 mg/kg/hr infusion postoperatively up to 24 hours) and oral memantine (5 mg BID [first week]; 10 mg BID [following three weeks]).
  Arms: NMDA active + Steroid active; NMDA active + Steroid placebo
Drug: Steroid active — Steroid active group will involve two doses of dexamethasone; 25 mg given prior to starting surgery and 25 mg given on the morning of second postoperative day.
  Arms: NMDA active + Steroid active; Steroid active + NMDA placebo
Drug: NMDA placebo — NMDA active group will involve normal saline (IV bolus pre-incision and infusion postoperatively up to 24 hours) and oral matching placebo to memantine (1 capsule BID [first week]; 1 capsule BID [following three weeks]).
  Arms: NMDA placebo + Steroid placebo; Steroid active + NMDA placebo
Drug: Steroid placebo — Steroid placebo group will involve two doses of normal saline; one dose given prior to starting surgery and one dose given on the morning of second postoperative day.
  Arms: NMDA active + Steroid placebo; NMDA placebo + Steroid placebo

SUMMARY:
The objective of the PAIN-STOP trial is to assess the feasibility of a larger randomized controlled trial (RCT) evaluating NMDA antagonists and IV steroids, as compared to placebo, in decreasing the chances of clinically significant persistent post-surgical pain (PPSP) after video assisted thoracoscopic surgeries (VATS). This is a multi-centre randomized, controlled clinical trial with a 2 x 2 factorial design. The pilot phase of the trial will recruit 48 patients and follow them for 3 months. Patients will be randomized to one of four groups: 1) NMDA active + Steroid placebo; 2) Steroid active + NMDA placebo; 3) NMDA active + Steroid active; 4) NMDA placebo + Steroid placebo.

DETAILED DESCRIPTION:
Persistent Post-Surgical Pain (PPSP) after Video Assisted Thoracic Surgery (VATS) lobectomy procedures is an important health problem for which there is no effective method of prevention. NMDA antagonists and steroids can modify pain signaling-sensitization pathways, and inflammatory-immune pathways, and hence can potentially prevent the development of PPSP. These agents have been safely used in thoracic surgeries to obtain many perioperative benefits, without increasing the harmful effects. Since these agents act by different biological mechanisms, it is appropriate to study their effects in a factorial design to increase the trial efficiency. Before conducting a large multicenter trial, we propose to establish the feasibility by carrying out this feasibility trial.

The objective of the PAIN-STOP trial is to assess the feasibility of a larger randomized controlled trial (RCT) evaluating NMDA antagonists and IV steroids, as compared to placebo, in decreasing the chances of clinically significant persistent post-surgical pain (PPSP) after video assisted thoracoscopic surgeries (VATS). This is a multi-centre randomized, controlled clinical trial with a 2 x 2 factorial design. The pilot phase of the trial will recruit 48 patients and follow them for 3 months. Patients will be randomized to one of four groups: 1) NMDA active + Steroid placebo; 2) Steroid active + NMDA placebo; 3) NMDA active + Steroid active; 4) NMDA placebo + Steroid placebo. Follow-up visit will be conducted in hospital; day 8 and month 2 by a phone call; and in person follow-up visits at 30 days and 3 months post-randomization; for patients who cannot attend in person, a telephone follow up will be done.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age,
* Planned elective VATS pulmonary lobectomy,
* Provide written informed consent to participate.

Exclusion Criteria:

* Current pain on the same side of the chest of moderate to severe intensity (>3/10 in 0-10 numerical rating scale (NRS) - where 0=no pain, 10=maximum pain),
* Known intracranial mass or cerebral aneurysm or raised intraocular pressure,
* Severe renal impairment (creatinine clearance based GFR of <30ml/min),
* Allergies to one or more of the study medications,
* Steroid treatment > 10mg/day of Prednisolone or its equivalent for > 3 weeks within the last 3 months,
* History of schizophrenia or bipolar disorder,
* History of drug addiction (prescription or non-prescription drug addiction diagnosed by a physician, excluding alcohol),
* Current diagnosis of Cushing's syndrome,
* Pregnancy,
* Previous participation in the PAIN-STOP trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Recruitment | 6 months
  Ability to recruit 90% of eligible patients.
Recruitment | 6 months
  Ability to recruit at least 4 patients per month per site, and complete the recruitment over a 6-month period.
Follow-up | 9 months
  Ability to obtain follow-up in >90% of enrolled patients, at three months.

SECONDARY OUTCOMES:
NRS - Incidence of PPSP | 3 months
  Intensity of PPSP on a scale of 0-10, at 3 months after randomization [0-10 numerical rating scale (NRS) - where 0=no pain, 10=maximum pain].
NRS - Incidence of PPSP with movement evoked | 3 months
  Incidence of PPSP (in and/or around the surgical scar) at 3 months after randomization, as the presence of movement evoked pain > 3/10 in 0-10 NRS.
Rate of change of postoperative pain intensity | 3 months
  The rate of change of postoperative pain intensity measured over time (pain trajectory).
Use of narcotic analgesic medication | 3 months
  Use of narcotic analgesic medication > 3 days/week beyond 4 weeks and up to 3 months after randomization.
Presence of NP | 3 months
  Presence of NP as > 3 out 7 items using DN4 scale, at measured at 3 months after randomization.
BPI score | 3 months
  Difference in interference with activities of daily living measured using Brief Pain Inventory interference score, measured at 3 months after randomization.
Thoracic surgery specific activity limitations | 3 months
  Difference in thoracic surgery specific activity limitations, measured at 3 months after randomization.
Change in global health status | 3 months
  Change in global health status measured using global impression of change (GIC) scale at 3 months after randomization.
Difference in Quality of Life | 3 months
  Difference in Quality of Life (QoL) using European Organization for Research and Treatment of Cancer (EORTC) QoL-30 at 3 months after randomization.

OTHER OUTCOMES:
Incidence of myocardial infarction and injury | 3 months
  Incidence of myocardial infarction and myocardial injury after noncardiac surgery (MINS)
Incidence of postoperative pneumonia | 3 months
  Incidence of postoperative pneumonia
Incidence of prolonged air-leak | 3 months
  Incidence of prolonged air-leak
Incidence of new intubation and positive pressure ventilation | 3 months
  Incidence of new intubation and positive pressure ventilation
Incidence of surgical site infection | 3 months
  Incidence of surgical site infection

CONTACTS AND LOCATIONS:
Overall Officials: PJ Devereaux, MD, PhD, Study Chair — McMaster University
Locations (2):
- Cleveland Clinic, Cleveland, Ohio, United States
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shanthanna H, Turan A, Vincent J, Saab R, Shargall Y, O'Hare T, Davis K, Fonguh S, Balasubramaniam K, Paul J, Gilron I, Kehlet H, Sessler DI, Bhandari M, Thabane L, Devereaux PJ. N-Methyl-D-Aspartate Antagonists and Steroids for the Prevention of Persisting Post-Surgical Pain After Thoracoscopic Surgeries: A Randomized Controlled, Factorial Design, International, Multicenter Pilot Trial. J Pain Res. 2020 Feb 12;13:377-387. doi: 10.2147/JPR.S237058. eCollection 2020. PMID 32104059